CLINICAL TRIAL: NCT03378388
Title: Effectiveness and Safety of Treatment With Vedolizumab in Adult Patients With Ulcerative Colitis or Crohn's Disease in Real Life
Brief Title: A Study to Assess the Effectiveness and Safety of Treatment With Vedolizumab in Adult Participants With Ulcerative Colitis (UC) or Crohn's Disease (CD) in Real Life
Acronym: GEVOL
Status: Terminated | Type: Observational
Why Stopped: Business Decision; Insufficient Enrollment
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vedolizumab-5039; U1111-1203-0268 (Registry Identifier: WHO)
Record Dates: First submitted 2017-12-11; First posted 2017-12-19 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases
Keywords: Drug therapy
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vedolizumab: Participants diagnosed with UC or CD, who fail or are intolerant to a previous biologic treatment or with contra-indication to anti-tumor necrosis factor alpha (TNF alpha) after failure of conventional treatments without exclusion except participant refusal, and were potentially eligible for a treatment with vedolizumab will be observed from the first prescription during consultation over a period of 24 months.

SUMMARY:
The purpose of this study is to describe in real life the effectiveness of treatment with vedolizumab.

DETAILED DESCRIPTION:
This is a prospective, non-interventional and pharmaco-epidemiological study of participants with IBD. The study will provide the real-life data of treatment effectiveness and safety of vedolizumab in adult participants with UC or CD.

The study will enroll approximately 300 participants. All participants will be enrolled in one observational group:

Vedolizumab

Data will be collected and observed for 24 months in the participants who will be freely chosen by physicians to prescribe vedolizumab at the end of consultation in the recruitment period.

This multi-center trial will be conducted in France. The overall time to participate in this study is 36 months, including participant's recruitment period of 12 months and treatment period of 24 months. Participants will make a minimum of 4 follow-up visits to the clinic in treatment period at Month 6, 12, 18, and 24.

ELIGIBILITY:
Inclusion Criteria:

1. Suffering from active disease of UC or CD according to the investigator's judgment.
2. In failure or intolerant to a previous biologic treatment, or with contra-indication to anti-TNFalpha after failure of conventional treatments, regardless of the line of treatment.
3. Meeting the same criteria as those described at the pre-screening.
4. Prescription of vedolizumab during consultation.
5. Able to be followed a priori over a period of 24 months.

Exclusion Criteria:

1. With exclusion criteria for vedolizumab and any contra-indication to vedolizumab: hypersensitivity to the active substance or to any of its excipients, active severe infections, such as tuberculosis, sepsis, cytomegalovirus, listeriosis, and opportunistic infections such as progressive multifocal leukoencephalopathy (PML).
2. Participation in an interventional study (but not in another non-interventional study).
3. Unclassified colitis.
4. Stomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who are biologically naive and are diagnosed with active disease of UC or CD according to investigator's judgement.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Complete Steroid-free Clinical Remission at Month 24 | Month 24
  Clinical remission is defined as Harvey Bradshaw-index (HBI) score less than or equal to (<=) 4 and partial mayo clinic score <=3. HBI score is used to measure disease activity of CD. It consists of clinical parameters: general well-being (0-4), abdominal pain (0-3), number of liquid stools per day, abdominal mass (0-3), and complications (score 1 per item). Total score is sum of individual parameters. Score ranges from minimum score of 0 to no pre-specified maximum score as it depends on number of liquid stools, where higher scores means more severe disease. Mayo score is an instrument designed to measure disease activity of UC and consists of 3 sub scores: stool frequency, rectal bleeding, and physician rating of disease activity, each graded from 0 to 3 with higher scores indicating more severe disease. These scores are summed to give a total score range of 0 to 9; where higher scores means more severe disease.

SECONDARY OUTCOMES:
Number of Participants with Complete Steroid-free Remission at Month 6, 12 and 18 | Months 6, 12, and 18
  Clinical remission is defined as HBI score <=4 and partial mayo clinic score <=3. HBI score is used to measure disease activity of CD. It consists of clinical parameters: general well-being (0-4), abdominal pain (0-3), number of liquid stools per day, abdominal mass (0-3), and complications (score 1 per item). Total score is sum of individual parameters. Score ranges from minimum score of 0 to no pre-specified maximum score as it depends on number of liquid stools, where higher scores means more severe disease. Mayo score is an instrument designed to measure disease activity of UC and consists of 3 sub scores: stool frequency, rectal bleeding, and physician rating of disease activity, each graded from 0 to 3 with higher scores indicating more severe disease. These scores are summed to give a total score range of 0 to 9; where higher scores means more severe disease.
Duration of Treatment in Participants Treated with Vedolizumab | Baseline up to Month 24
Number of Participants who had Treatment Failure When Treated With Vedolizumab | Baseline up to Month 24
Number of Treatment Lines in Participants Treated with Vedolizumab | Baseline up to Month 24
Number of Naïve Participants Ineligible to Anti TNF Alpha | Baseline up to Month 24
Number of Non-naïve Participants Ineligible to Anti TNF Alpha | Baseline up to Month 24
Number of Participants who Experience at Least one Treatment-emergent Adverse Event (TEAE) | Baseline up to Month 24
Number of Participants with Non-serious Adverse Drug Reactions (ADRs) | Baseline up to Month 24
Number of Participants with Special Situation Report (SSR) | Baseline up to Month 24
Number of Participants with Product Quality Issues | Baseline up to Month 24
  A product quality issue refers to defects related to the safety, identity, strength, quality, or purity of the product or with the physical characteristics, packaging, labelling, or design of the product.
Number of Participants with Markedly Abnormal Laboratory Values | Baseline up to Month 24
Patient Reported Outcomes (PRO) 1: Quality of Life | Months 6, 12, 18 and 24
  Participant's Quality of Life (PRO-1) will be measured by the inflammatory bowel disease questionnaire (IBDQ). The IBDQ is a 32-item questionnaire that measures 4 dimensions: bowel symptoms (10 items), emotional disorders (12 items), systemic symptoms (5 items), and social function (5 items). Each item is measured according to the Likert technique. Within dimensions, each question presents seven possible answers/points. Each domain score is the sum of 8 responses each ranging from 1 to 7, where 1 indicates worst function and 7 the best. The sub-score ranges from 8 to 56; a higher score indicating a better quality of life. Hence, the total score ranges from 32 to 224, with higher scores representing better quality of life.
PRO 2: Number of Participants who met Item 1 and 2 on the Partial Mayo Score and Item 2 and 3 on the HBI | Months 6, 12, 18 and 24
Number of Participants With Concordance Between PRO-2 and Physicians Answers | Baseline up to 24 Months
Number of Participants who had Relapses | Baseline up to Month 24
  Number of participants with relapses will be collected through hospital reports which will be provided by the investigator.
Number of Participants who had Surgery | Baseline up to Month 24
  Number of participants with surgery will be collected through hospital reports which will be provided by the investigator.
Number of Participants who had Complications due to Adverse Events (AEs) | Baseline up to Month 24
Number of Participants who had Hospitalizations | Baseline up to Month 24
  Number of participants with hospitalizations will be collected through hospital reports which will be provided by the investigator.
Number of Participants who had Absenteeism | Baseline up to Month 24
  Number of participants with absenteeism will be collected by the participants using a self-administered questionnaire.
Number of Participants with Vedolizumab Effectiveness on Extra-intestinal Manifestations or Fistula | Baseline up to Month 24
  Number of participants who had effectiveness of vedolizumab on extra-intestinal manifestations or fistula will be assessed. Extra-intestinal manifestations of pathology such as skin, articular, ocular, metabolic, bone, hepato-pancreato-biliary, neurological, cardiovascular diseases and complications related to anal fistula is planned to be assessed.
Number of Participants with Mucosal Healing Having Undergone Endoscopy | Months 6, 12, 18 and 24
  Mucosal healing is defined either as the absence of any ulcer (Crohn's Disease Endoscopic Index of Severity [CDEIS] at 0) for CD participants and as a Mayo clinic endoscopic subscore <=1 for UC participants.
Percentage of Physicians Following the French National Consensus for the Management of IBD into Clinical Practice | Baseline up to Month 24
  Percentage of physicians following the French national consensus for the management of IBD into clinical practice.
Number of Participants with Comorbodities, Previous Line of Therapy and Concomitant Treatments | Baseline up to Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (13):
- France (13):
  - Centre Hospitalier Cote Basque, Bayonne
  - Ch de Blois, Blois
  - Clinique du palais, Grasse
  - Ghef Ch Marne La Vallee, Jossigny
  - Ctre Hosp St Joseph Et St Luc, Lyon
  - Hopital Edouard Herriot, Lyon
  - Hopital Saint Eloi-Chru Montpellier, Montpellier
  - Ch Lyon Sud, Pierre-Bénite
  - Polyclinique Cote Basque Sud, Saint-Jean-de-Luz
  - HOPITAL NORD-CHU de SAINT-ETIENNE, Saint-Priest-en-Jarez
  - Clinique Ambroise Pare, Toulouse
  - HOPITAUX DE BRABOIS-CHRU de NANCY, Vandœuvre-lès-Nancy
  - Gh mutualiste les portes du sud, Vénissieux

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/